CLINICAL TRIAL: NCT06968234
Title: Exploring Clinical Characteristics of Liver Disease Patients Based on Digestive Metabolic Exhaled Air
Status: Recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B2025-179R
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Cirrhosis; Microbiota; Breath Tests
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- H₂ abnormality: Fasting end-expiratory H₂ ≥ 10 ppm, indicating excessive growth of hydrogen-producing bacteria in the gut.
- CH₄ abnormality: Fasting end-expiratory CH₄ ≥ 5 ppm, indicating excessive growth of methanogenic archaea in the gut.
- H₂S abnormality: Fasting end-expiratory H₂S ≥ 50 ppb, indicating excessive growth of hydrogen sulfide-producing bacteria in the gut.
- NO abnormality: Fasting end-expiratory NO ≥ 15 ppb, indicating the presence of low-grade intestinal inflammation or eosinophilic inflammation.
- Small Intestinal Bacterial Overgrowth (SIBO): Defined as end-expiratory H₂ ≥ 10 ppm or CH₄ ≥ 5 ppm.

SUMMARY:
Cirrhosis is a common digestive system disease and represents the final stage of the progression of various chronic liver diseases. During cirrhosis, the intestinal microenvironment is affected due to liver damage and increased portal venous pressure. Displacement of gut microbiota is closely related to the occurrence and development of cirrhosis. Disruption of the gut microbiota is associated with changes in the levels of nitric oxide (NO), hydrogen (H₂), methane (CH₄), and hydrogen sulfide (H₂S). Breath testing is an emerging method for assessing gut microbiota. This project aims to investigate the characteristics and prognosis of patients with chronic liver disease by detecting exhaled breath markers such as nitric oxide (NO), hydrogen (H₂), methane (CH₄), and hydrogen sulfide (H₂S), in conjunction with results from serological tests, gut microbiota analysis, and radiomics. The goal is to identify new diagnostic biomarkers and therapeutic targets, to recognize high-risk patients at an early stage, and to improve patient survival rates and quality of life.

ELIGIBILITY:
Inclusion Criteria:

① Patients diagnosed with chronic liver disease or cirrhosis through liver biopsy pathology or clinical laboratory and imaging examinations;

② Undergo molecular breath testing within one week of admission.

Exclusion Criteria:

* Patients who have received antibiotic treatment within one month; ② Patients with severe pulmonary diseases, such as chronic obstructive pulmonary disease (COPD), asthma, or lung malignancies that have not been clinically cured; ③ Patients who are unable to successfully complete the molecular breath test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic liver disease and cirrhosis hospitalized at Fudan University Affiliated Zhongshan Hospital, Shanghai Institute of Geriatric Medicine, and Minhang District Central Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal bleeding | 2 months
  Defined as a decrease in hemoglobin by 2 g/L or the presence of active bleeding, hematochezia, or other signs of bleeding.

SECONDARY OUTCOMES:
The occurrence of clinical events | 6 months, 1 year, and 2 years
  The occurrence of events such as gastrointestinal bleeding, ascites progression, overt jaundice, and portal vein thrombosis at 6 months, 1 year, and 2 years, as well as the incidence of liver cancer, liver transplantation, or survival and death.

CONTACTS AND LOCATIONS:
Overall Officials: Shiyao Chen, Ph.D., Principal Investigator — Shanghai Zhongshan Hospital
Locations (3):
- China (3):
  - Shanghai Geriatrics Medical Center, Shanghai, Shanghai Municipality
  - Shanghai Minhang District Central Hospital, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Shanghai, Shanghai Municipality